CLINICAL TRIAL: NCT04048421
Title: A Phase II Study to Evaluate the Feasibility and Safety of Hybrid Transvaginal Natural Orifice Transluminal Endoscopic Surgery for Treatment of Patients With Colon Cancer
Brief Title: Feasibility and Safety of Hybrid Transvaginal Natural Orifice Transluminal Endoscopic Surgery for Colon Cancer
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Renmin Hospital of Wuhan University (Other)
Responsible Party: Principal Investigator, Tao Fu, Chief of Department of Gastrointestinal Surgery II, Renmin Hospital of Wuhan University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: vNOTESCA
Record Dates: First submitted 2019-07-03; First posted 2019-08-07 (Actual); Last update posted 2023-08-03 (Actual); Status verified 2023-08

CONDITIONS: Colon Cancer; Natural Orifice Transluminal Endoscopic Surgery
MeSH Terms: conditions — Colonic Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- hvNOTES group (Experimental): Participants will undergo hvNOTES radical colectomy.
  Interventions: Procedure: hvNOTES radical colectomy

INTERVENTIONS:
Procedure: hvNOTES radical colectomy — With the patient under general anesthesia, pneumoperitoneum is achieved. Three trocars are inserted, one 12 mm or 5 mm in the umbilicus and two 5 mm in the right and/or left flanks. Mobilization of the splenic flexure or the hepatic flexure is performed with an initial traditional laparoscopic approach. A single-port is inserted into the abdominal cavity transvaginally through the colpotomy. Then most of the procedures are performed transvaginally with conventional rigid laparoscopic instruments. The corresponding arteries and veins are divided. The mesocolon is mobilized. The small intestine/colon/rectum are then divided with stapler. The specimen is removed transvaginally. Intracorporeal anastomosis is performed as per the surgeon's standard of care. For sigmoidectomy, the colon is then exteriorized and the anvil is fixed in the colon. An end-to-end anastomosis is performed using a circular stapler. Drainage tubes may be used.

SUMMARY:
This study aims to evaluate the safety and efficacy of radical colectomy with hybrid transvaginal natural orifice transluminal endoscopic surgery (hvNOTES). This is a prospective, single-arm, multicenter, uncontrolled, open-label phase II study in 55 eligible subjects with resectable colon cancer. After informed consent, patients will be sent to have hvNOTES radical colectomy by surgeons with good experience in laparoscopic colorectal surgery. Patients' demographic, operative detail and postoperative outcomes including conversion to open surgery, operating time, blood loss, pain score, resumption of gastrointestinal function, postoperative complications, length of hospital stay, sexual function, quality of recovery, recurrence rate, recurrence patterns, relapse-free survival, and overall survival will be recorded prospectively. The results of the patients will be assessed to validate safety, functional outcomes or oncologic outcomes of hvNOTES colectomy.

ELIGIBILITY:
Inclusion Criteria:

1. Female.
2. Age: over 18 and below 80 years old.
3. BMI < 28 kg/m^2.
4. American Society of Anesthesiologists score of class I to III.
5. Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1.
6. Colonic adenocarcinoma by endoscopy with biopsy.
7. Tumor size ≤ 5 cm.
8. Involving a single colon segment:

   1. Right colon from the ileocecal valve up to and including the hepatic flexure.
   2. Left colon from the splenic flexure to the junction of the sigmoid and descending colon.
   3. Sigmoid colon between the descending colon and the rectum (at least 15 cm from the dentate).
9. Clinical stage cT1, T2, or T3, cN0, N1, N2.
10. No advanced local disease that renders laparoscopic resection impossible.
11. No transverse colon cancer (between distal hepatic flexure and proximal splenic flexure).
12. No distant metastasis in preoperative studies.
13. Complete preoperative colonoscopy demonstrating no synchronous colon cancers.
14. Require one of the following elective operations that may be safely performed by current techniques:

    1. Right hemicolectomy
    2. Left hemicolectomy
    3. Subtotal colectomy
    4. Sigmoid colectomy
15. Patients who agree with participating in the clinical study with informed consents. And with willingness and ability to comply with the requirements of the study protocol including follow-up.

Exclusion Criteria:

1. Patients who have never experienced complete sexual intercourse before the operation.
2. Previous intestinal surgery with any cause.
3. cT4 tumor.
4. Complications of colon cancer (bleeding, obstruction, or perforation).
5. Previous neoadjuvant chemotherapy or radiotherapy for colon cancer.
6. Patients who are diagnosed with other malignancies within 5 years.
7. Vulnerable patients.
8. Vaginal stenosis.
9. Prior reconstructive surgery of the vagina not including hysterectomy.
10. Unstable angina or myocardial infarction within the past 6 months.
11. Cerebrovascular accident within the past 6 months.
12. Continuous systemic steroid therapy within 1 month before the surgery.
13. Patients who participating or participated in other clinical trial within 6 months.
14. Pregnancy or breastfeeding.
15. Any history of pelvic radiation.
16. Anticipated need for an ostomy at the time of operation.
17. Patients requiring urgent or emergent surgery.
18. Patients with prior or suspected diagnosis of inflammatory bowel disease such as Crohn's disease, ulcerative colitis, or familial polyposis.

Ages: 18 Years to 80 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 55 (Estimated)
Dates: Start 2019-12-20 (Actual); Primary Completion 2024-11-30 (Estimated); Study Completion 2025-11-30 (Estimated)

PRIMARY OUTCOMES:
Postoperative complications | up to 90 days after surgery
  The primary end point is major complication during surgery or within 90 days after surgery. A major intraoperative and postoperative complication is defined as a surgical or medical complication with a CTCAE grade of III or higher. The most severe complication in a patient was considered for the classification of the primary end point.

SECONDARY OUTCOMES:
Conversion to laparoscopic or open surgery | during the surgery
  One of the secondary outcome measures is the rate of conversion to laparoscopic or open surgery as an indicator of surgical technical difficulty. Conversion is defined as the use of a laparoscopic port for the anastomosis, or a laparotomy wound for any part of the mesocolon dissection or the anastomosis.
Concentration of c-reactive protein (CRP) | 1 and 3 postoperative days
  C-Reactive Protein (CRP) values on postoperative day 1and 3.
Concentration of procalcitonine (PCT) | 1 and 3 postoperative days
  Procalcitonine (PCT) values on postoperative day 1and 3.
Complete pathological assessment of CME specimens | up to 1 week after surgery
  Complete mesocolic excision (CME) is defined as complete resection of the mesocolon with its anatomical envelope. Rate of complete and near-CME achieved with hvNOTES, based on standard pathologic assessment of CME specimens.
Postoperative pain assessed by the numeric rating scale (NRS) | up to 1 week after surgery
  Pain score assessments: The investigator's staff will provide a rating scale to the patients to self-rate and record their pain at baseline (prior to surgery), at 24, 48, 72, 96, 120, 144, and 168 hours following the procedure end time (or discharge if earlier) postoperatively using the numeric rating scale (NRS) where 0 is for no pain and 10 is for the worst pain imaginable.
Amount of narcotic pain medication administered | up to 1 week after surgery
  The amount of narcotic pain medication administered through postoperative day 7 (or discharge if earlier) will be recorded (total dose of morphine equivalent during hospitalization and average dose per day).
Time to first flatus after surgery | up to 1 week after surgery
  Time to first flatus is defined as days from a colectomy procedure to first occurrence of flatus during subject's postoperative recovery.
Number of harvested lymph nodes | up to 1 week after surgery
  Number of harvested Lymph nodes according to the pathological report.
R0 resection | up to 1 week after surgery
  Rate of resection without any affected margins during the surgical procedure according to the pathological report.
Length of hospital stay | up to 4 weeks after surgery
  Days in the hospital after surgery.
Sexual function assessment | baseline, 6 months, and 12 months after surgery
  Patient self-reported sexual functions as assessed by the Female Sexual Function Index (FSFI). The FSFI is a 19-item questionnaire to rate sexual function between 2.0 and 36.0, where 2.0 is low sexual function and 36.0 is high sexual function.
Quality of recovery: Quality of Recovery 40 questionnaire (QoR-40) | 14 days after surgery
  Patient's quality of recovery is assessed by using the Quality of Recovery 40 questionnaire (QoR-40, score range: 40-200). Higher values represent better outcomes. The validate questionnaire measure quality of recovery by evaluating patients' comfort, emotions, physical independence, and support using the same scale.
Satisfaction with surgical scars: Validated questionnaire Patient Scar Assessment Questionnaire (PSAQ) | 3, 6, and 12 months after surgery
  Validated questionnaire Patient Scar Assessment Questionnaire (PSAQ, score range: 28-102) will be administered to assess the patient's perception of scarring. Lower values represent better outcomes. The PSAQ consists of 5 subscales: Appearance, symptoms, consciousness, satisfaction with appearance, and satisfaction with symptoms.
Quality of Life Questionnaire (QLQ) of the European Organisation for Research and Treatment of Cancer (EORTC) QLQ-C30 | baseline, 3 and 12 months after surgery
  Quality of Life Questionnaire (QLQ) of the European Organisation for Research and Treatment of Cancer (EORTC) QLQ-C30 Score 3 months and 1 year after the procedure. This scale has functional, global health, and symptoms subscales/items all scored from 0 to 100. Higher scores on these subscales indicate high level of functioning, high quality of life, and high level of symptomatology, respectively.
Postoperative recurrence patterns | 2 years after surgery
  The recurrence patterns are determined according to the primary recurrence site diagnosed radiologically (CT, US, MRI, or PET-CT), or with histologic proof (ascitic cytology, colonoscopic biopsy, or surgery).
Relapse-free survival | 2 years after surgery
  Relapse-free survival is defined as the time from random assignment until disease relapse or death from any cause.
Overall survival | 2 years after surgery
  Overall survival is defined as time from surgery to death.

CONTACTS AND LOCATIONS:
Overall Officials: Tao Fu, MD, Principal Investigator — Wuhan University Renmin Hospital
Locations (6):
- China (6):
  - Beijing Friendship Hospital of Capital Medical University, Beijing, Beijing Municipality
  - Daping Hospital of Army Medical University, Chongqing, Chongqing Municipality
  - Renmin Hospital of Wuhan University, Wuhan, Hubei
  - The Third Xiangya Hospital of Central South University, Changsha, Hunan
  - Qingdao Municipal Hospital, Qingdao, Shandong
  - The Second Affiliated Hospital of Zhejiang University, Hangzhou, Zhejiang

IPD SHARING:
Plan to Share IPD: Yes
Data obtained through this study may be provided to qualified researchers with academic interest in natural orifice transluminal endoscopic surgery. Data or samples shared will be coded, with no protected health information (PHI) included. Approval of the request and execution of all applicable agreements (i.e. a material transfer agreement) are prerequisites to the sharing of data with the requesting party.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Data requests can be submitted starting 9 months after article publication and the data will be made accessible for up to 24 months. Extensions will be considered on a case-by-case basis.
Access Criteria: Access to trial IPD can be requested by qualified researchers engaging in independent scientific research, and will be provided following review and approval of a research proposal and Statistical Analysis Plan (SAP) and execution of a Data Sharing Agreement (DSA). For more information or to submit a request, please contact tfu001@whu.edu.cn.

REFERENCES:
- [Background] Rattner D, Kalloo A; ASGE/SAGES Working Group. ASGE/SAGES Working Group on Natural Orifice Translumenal Endoscopic Surgery. October 2005. Surg Endosc. 2006 Feb;20(2):329-33. doi: 10.1007/s00464-005-3006-0. No abstract available. PMID 16402290
- [Background] Rattner DW, Hawes R, Schwaitzberg S, Kochman M, Swanstrom L. The Second SAGES/ASGE White Paper on natural orifice transluminal endoscopic surgery: 5 years of progress. Surg Endosc. 2011 Aug;25(8):2441-8. doi: 10.1007/s00464-011-1605-5. Epub 2011 Feb 27. No abstract available. PMID 21359881
- [Background] Moloney JM, Gan PS. Hybrid Transvaginal NOTES and Mini-Laparoscopic Colectomy: Benefit Through Synergy. JSLS. 2016 Oct-Dec;20(4):e2016.00062. doi: 10.4293/JSLS.2016.00062. PMID 27904307
- [Background] Lamm SH, Zerz A, Efeoglou A, Steinemann DC. Transrectal Rigid-Hybrid Natural Orifice Translumenal Endoscopic Sigmoidectomy for Diverticular Disease: A Prospective Cohort Study. J Am Coll Surg. 2015 Oct;221(4):789-97. doi: 10.1016/j.jamcollsurg.2015.07.012. Epub 2015 Jul 21. PMID 26282488
- [Background] Bulian DR, Runkel N, Burghardt J, Lamade W, Butters M, Utech M, Thon KP, Lefering R, Heiss MM, Buhr HJ, Lehmann KS. Natural Orifice Transluminal Endoscopic Surgery (NOTES) for colon resections--analysis of the first 139 patients of the German NOTES Registry (GNR). Int J Colorectal Dis. 2014 Jul;29(7):853-61. doi: 10.1007/s00384-014-1883-1. Epub 2014 May 7. PMID 24798629
- [Background] D'Hondt M, Devriendt D, Van Rooy F, Vansteenkiste F, Dozois E. Transvaginal pure NOTES sigmoid resection using a single port device. Tech Coloproctol. 2014 Jan;18(1):77-80. doi: 10.1007/s10151-013-1005-z. Epub 2013 Apr 6. PMID 23564271
- [Background] Alba Mesa F, Amaya Cortijo A, Romero Fernandez JM, Komorowski AL, Sanchez Hurtado MA, Fernandez Ortega E, Sanchez Margallo FM. Transvaginal sigmoid cancer resection: first case with 12 months of follow-up--technique description. J Laparoendosc Adv Surg Tech A. 2012 Jul-Aug;22(6):587-90. doi: 10.1089/lap.2011.0469. Epub 2012 Jun 12. PMID 22690651
- [Background] Alba Mesa F, Amaya Cortijo A, Romero Fernandez JM, Komorowski AL, Sanchez Hurtado MA, Sanchez Margallo FM. Totally transvaginal resection of the descending colon in an experimental model. Surg Endosc. 2012 Mar;26(3):877-81. doi: 10.1007/s00464-011-1919-3. Epub 2011 Sep 23. PMID 21947741
- [Background] Lacy AM, Delgado S, Rojas OA, Almenara R, Blasi A, Llach J. MA-NOS radical sigmoidectomy: report of a transvaginal resection in the human. Surg Endosc. 2008 Jul;22(7):1717-23. doi: 10.1007/s00464-008-9956-2. Epub 2008 May 7. PMID 18461385
- [Background] Sodergren MH, Clark J, Athanasiou T, Teare J, Yang GZ, Darzi A. Natural orifice translumenal endoscopic surgery: critical appraisal of applications in clinical practice. Surg Endosc. 2009 Apr;23(4):680-7. doi: 10.1007/s00464-008-0278-1. Epub 2009 Jan 1. PMID 19118425
- [Background] Whiteford MH, Spaun GO. A colorectal surgeons viewpoint on natural orifice translumenal endoscopic surgery. Minerva Chir. 2008 Oct;63(5):385-8. PMID 18923349
- [Background] Park JS, Choi GS, Lim KH, Jang YS, Kim HJ, Park SY, Jun SH. Clinical outcome of laparoscopic right hemicolectomy with transvaginal resection, anastomosis, and retrieval of specimen. Dis Colon Rectum. 2010 Nov;53(11):1473-9. doi: 10.1007/DCR.0b013e3181f1cc17. PMID 20940594
- [Background] Alba Mesa F, Sanchez Hurtado MA, Sanchez Margallo FM, Romero Fernandez JM, Amaya Cortijo A, Fernandez Ortega E, Komorowski AL. Laparoscopy-assisted transvaginal resection of sigmoid cancer. Eur J Surg Oncol. 2014 Jun;40(6):713-8. doi: 10.1016/j.ejso.2014.01.008. Epub 2014 Feb 7. PMID 24560464
- [Background] Noguera JF, Cuadrado A, Dolz C, Olea JM, Garcia JC. Prospective randomized clinical trial comparing laparoscopic cholecystectomy and hybrid natural orifice transluminal endoscopic surgery (NOTES) (NCT00835250). Surg Endosc. 2012 Dec;26(12):3435-41. doi: 10.1007/s00464-012-2359-4. Epub 2012 May 31. PMID 22648123
- [Derived] Fu T, Ren J, Yao H, Huang B, Sun L, Li X, Tong W. Feasibility and safety of hybrid transvaginal natural orifice transluminal endoscopic surgery for colon cancer: Protocol for a multicenter, single-arm, phase II trial (vNOTESCA). Heliyon. 2023 Sep 23;9(10):e20187. doi: 10.1016/j.heliyon.2023.e20187. eCollection 2023 Oct. PMID 37780770

DOCUMENTS (1):
  • Informed Consent Form (2022-06-16): https://cdn.clinicaltrials.gov/large-docs/21/NCT04048421/ICF_001.pdf